CLINICAL TRIAL: NCT00110825
Title: Behavioral Maintenance Treatment for Smoking Cessation
Brief Title: Behavioral Smoking Cessation Treatment - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Professor Joel D Killen, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-17441-1; R01-DA17441-1; DPMCDA; R01DA017441 (NIH)
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-06

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — extended treatment with cognitive behavior therapy

SUMMARY:
Our primary goal is to examine the effectiveness of a multi-factor maintenance treatment strategy in promoting longer-term smoking abstinence. We will also conduct secondary analyses of mediators and moderators of treatment response.

DETAILED DESCRIPTION:
400 adult smokers will be randomized. Our primary goal is to examine the effectiveness of a multi-factor maintenance treatment strategy in promoting longer-term smoking abstinence. All smokers will receive the same "Acute Phase Treatment" that combines nicotine patch, bupropion and intensive self-regulatory skills training. Nicotine patches will be provided for 8 weeks and bupropion and skills training will be provided for of 9 weeks. Participants will then enter a "Maintenance Treatment Phase" during which half (n=200) will receive three individualized relapse prevention training sessions spread over a 12 week period. They will also receive 12 weeks of self-administered RPT administered via written treatment modules. Finally, telephone counseling will be provided in conjunction with an Interactive Voice Response system (IVR) that will allow early detection of smoking "slips" and rapid response by treatment staff. The other half (n=200) will be assigned to a control condition that consists of three counselor-led sessions of "supportive therapy" spread over a 12 week period. P

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult cigarette smokers smoking at least 10 cigarettes per day

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding
* Currently diagnosed with a seizure disorder, major depression, liver disease, kidney disease, congestive heart failure
* History of a seizure, seizure disorder, significant head trauma or central nervous system tumor
* Family history of seizures
* Currently using intravenous drugs
* Currently using any drugs (marijuana, alcohol, cocaine, opiates, stimulants, etc.) on a daily basis
* Currently using any over-the-counter stimulants and anorectics (diet pills)
* Currently on bupropion (Wellbutrin, Wellbutrin SR) or other antidepressants, monoamine oxidase inhibitors, antipsychotics, benzodiazepines, theophylline, systemic steroids or levodopa
* Currently on NRT or bupropion (Zyban)
* Current or past diagnosis of anorexia nervosa or bulimia nervosa
* Previous allergic response to bupropion or NRT
* Previous failed quit attempt using NRT and bupropion in combination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of cigarette abstinence | 8 weeks, 20 weeks, 52 weeks

SECONDARY OUTCOMES:
Analog mood scales | 8 weeks, 20 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Killen, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Stop Smoking Program, San Jose, California, United States

REFERENCES:
- [Result] Killen JD, Fortmann SP, Schatzberg AF, Arredondo C, Murphy G, Hayward C, Celio M, Cromp D, Fong D, Pandurangi M. Extended cognitive behavior therapy for cigarette smoking cessation. Addiction. 2008 Aug;103(8):1381-90. doi: 10.1111/j.1360-0443.2008.02273.x. PMID 18855829